CLINICAL TRIAL: NCT07341204
Title: Improvement of Sustained Attention Through Immersive Virtual Reality in Neurodivergent Children
Brief Title: How Virtual Reality Can Help Neurodivergent Children Improve Their Attention
Acronym: Attend-VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYIT IRB-2026-367
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Autism; Autism Disorder; ADHD - Attention Deficit Disorder With Hyperactivity; Attention Deficit Disorder
Keywords: attention; impulsivity; distractability; focus; VR; Immersive Virtual Reality
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine the impact of the VR game (Electrical Maze) on sustained attention outcomes in children with Neurodivergent conditions (ASD, ADHD, SLD, and DCD). The usage of an active intervention classifies this study as an interventional design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Does participation in a 6-week VR-based program improve attentional skills in neurodiverse children? (Experimental): The research design comprises a nonequivalent quasi-experimental, multi-group pre- and post-test design (neurodivergent and neurotypical). The pre-test and post-test will consist of the Test of Variables of Attention (TOVA) and the RightEye assessment. These measures will be administered at the clinical site (ISF). The intervention consists of two 25-minute VR sessions per week for 6 weeks.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — Participants will engage in an immersive virtual reality (VR) game intervention designed to improve visual attention skills. The intervention employs a VR game called Electrical Maze, which requires players to maintain sustained visual attention and respond to game challenges that develop focus and inhibitory control.
  Each participant will complete scheduled VR gaming sessions that target attentional skill development. During the sessions, children interact with the Electrical Maze game, which presents visual tasks that require them to identify and respond to specific visual cues while inhibiting responses to non-target stimuli.

SUMMARY:
The goal of this study is to determine whether playing a virtual reality (VR) game can help neurodivergent children pay attention for extended periods. The study includes children ages 9 to 18 who have autism, ADHD, learning differences, or movement coordination challenges. The program lasts for 6 weeks. During this period, children will play a VR game twice per week, with each session lasting 25 minutes.

DETAILED DESCRIPTION:
The purpose of this quasi-experimental study is to investigate the impact of an immersive virtual reality (VR) game intervention on sustained attention in neurodivergent children aged 9 to 18 years. This project aligns with previous study dosages designed as a 6-week program targeting children diagnosed with autism spectrum disorder (ASD), attention-deficit/hyperactivity disorder (ADHD), specific learning disorder (SLD), or developmental coordination disorder (DCD) (neurodivergent disorders). Participants will be recruited through convenience sampling in the local community and will participate in two 25-minute VR sessions per week for 6 weeks.

This study examines the effectiveness of a VR-based attention-training program by comparing pre- and post-intervention data using the Test of Variables of Attention (TOVA) and the Right Eye assessment. Repeated-measures ANOVA will be used to evaluate changes in sustained attention, including omission rates and response times. The findings will provide insight into how immersive VR games can enhance attention and engagement in daily activities among neurodivergent children, thereby facilitating the integration of technology-based interventions into therapeutic practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ASD, ADHD, SLD, or DCD confirmed by a licensed clinician or documented in medical/educational records (DSM-5 or equivalent).
* Parent/guardian consent and participant assent (age-appropriate).
* Ability to follow simple verbal instructions and to participate in 25-minute VR sessions twice weekly for 6 weeks.
* Stable medication regimen for attention- or behavior-related medications for ≥4 weeks prior to baseline (or not taking such medications).
* Visual and auditory ability adequate for VR tasks (with or without usual corrective lenses/hearing aids).
* Availability to attend all scheduled sessions at the clinical site across the 6-week period.

Exclusion Criteria:

* History of photosensitive epilepsy or any uncontrolled seizure disorder.
* Severe intellectual disability or severe communication impairment that prevents understanding/participation (e.g., non-responsive to simple commands required by the VR tasks).
* Severe visual, auditory, or motor impairment that prevents safe or functional use of the VR system (e.g., inability to hold controllers or view the headset even with correction).
* Recent (within 6 months) significant brain injury or neurosurgery. Significant history of motion sickness, severe vestibular disorder, or prior intolerance to immersive VR.
* Any medical or implanted device contraindicated for VR/headset use (if applicable).

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
RightEye Assessment: | Individual tests: 60 seconds (e.g., saccades) to 4-5 minutes (e.g., reaction time or pursuit tasks). Total session: 15-20 minutes, including 1-2 minutes for 9-point calibration and setup.
  The RightEye system uses an infrared camera-based sensor bar attached to a monitor to objectively measure and analyze eye movements in real-time. It quantifies changes in attention-related oculomotor functions, including saccadic accuracy, smooth pursuit, reaction time, distractibility, and sustained attention. These metrics provide objective biomarkers for inattention and impulsivity, supporting occupational therapy goals of enhancing visual-motor integration, executive function, and participation in daily activities like reading or classroom engagement.
Test of Variables of Attention (TOVA) | Standard visual test: 21.6 minutes (4 quarters of 5.4 minutes). Full session: 30-45 minutes (setup/review); short form for younger children (10.8 minutes; used for ages 9+).
  The TOVA objectively measures sustained attention and inhibitory control via responses to visual stimuli (targets vs. non-targets). In this study, the visual TOVA will assess pre- and post-VR changes in attention in children with neurodevelopmental conditions, targeting omission errors, commission errors, response time, and response time variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Inclusive Sports and Fitness, Inc., Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No